CLINICAL TRIAL: NCT06291662
Title: Evaluation of Performance Characteristics and Applicability in Oncology of Devices Customized Medical Devices Made by 3D Printing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kathleen McGreevy (Other)
Responsible Party: Sponsor-Investigator, Kathleen McGreevy, Chief Operating Officer, Meyer Children's Research Institute, Meyer Children's Hospital IRCCS
Organization: Meyer Children's Hospital IRCCS (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRECISE_IC
Record Dates: First submitted 2024-02-19; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Sarcoma; Intracranial Neoplasm; Pelvic Bone Neoplasm
MeSH Terms: conditions — Sarcoma; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Oncologic patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pelvic bone neoplasm (Experimental): Patients with primary tumor of the pelvic bone; Primary meta-diaphysial tumor of the long bones; squamous cell carcinoma of the oral cavity involving the maxillary upper and/or lower.
  Interventions: Device: 3D printer applications
- Sarcoma pediatric patients (Experimental): Patients with primary sarcoma of bone and soft parts involving the scapula, the pelvis and upper and lower limbs; brain tumor.
  Interventions: Device: 3D printer applications
- Intracranial oncologic pathology (Experimental): Patients with intracranial oncologic pathology with bone involvement and lesions of the skull theca primary or secondary.
  Interventions: Device: 3D printer applications

INTERVENTIONS:
Device: 3D printer applications — Patients will undergo TC/MRI as per routinary care. Custom 3D-devices will be printed on the basis of these images. The device will be used to establish pre-operative surgical options in terms of tissue/bones demolition/reconstruction.

SUMMARY:
Technologies 3D are demonstrating enormous potential for innovation in the field of surgery,introducing the concept of "treatment customization" (from planning surgery to implant design and manufacturing) on the patient's anatomy, simply by taking advantage of the patient's own common diagnostic images and the flexibility of 3D printing. In fact, this new construction technology allows the construction of the complex anatomical geometries with economy, simplicity and on scales of production unattainable by other traditional technologies. This new construction technology allows, in fact, the construction of complex anatomical geometries with economy, simplicity and on scales of production unattainable by other traditional technologies.

ELIGIBILITY:
Inclusion Criteria:

* Primary tumor of the pelvic bone Primary meta-diaphysial tumor of the long bones; squamous cell carcinoma of the oral cavity in the upper and/or lower jaw. over 10 years of age
* Primary sarcoma of bone and soft parts involving the scapula, the pelvis and upper and lower limbs; brain tumor aged 7-18 years
* Intracranial oncologic pathology with bone involvement and lesions of the skull theca primary or secondary aged 18-70years
* signed informed consent form

Exclusion Criteria:

* inoperability;
* presence of pathological fractures.

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
3D model feasibility for pre-surgical making decisions | through study completion, an average of 1 year
  Number of cases in which the time interval between prescription and delivery of the device exceeds 20 days
Surgical time | through study completion, an average of 1 year
  Number of procedures in which the surgical outcome can be considered optimal (taking planning as a reference) by comparing CT images and evaluating the margins at final histologic analysis.
Device feasibility | through study completion, an average of 1 year
  Proportion of failed surgeries due to a positive or contaminated finding of the margin of bone resection on final histological examination. verified by comparing the expected outcome (i.e., planning output) and the actual outcome (on the postoperative CT scan).

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Azienda Ospedaliero-Universitaria Careggi (AOUC), Florence
  - Meyer Children's Hospital IRCCS, Florence
  - Azienda Ospedaliero Universitaria Senese (AOUS), Siena

IPD SHARING:
Plan to Share IPD: No